CLINICAL TRIAL: NCT00961415
Title: Open-label Study of Bevacizumab Maintenance Therapy (AVASTIN®) With or Without Pemetrexed After First-line Chemotherapy With Bevacizumab-cisplatin-pemetrexed in Patients With Advanced, Metastatic or Recurrent Non-squamous Non-small Cell Lung Cancer (NSCLC)
Brief Title: AVAPERL1 Study: A Study of Avastin (Bevacizumab) With or Without Pemetrexed as Maintenance Therapy After Avastin in First Line in Patients With Non-Squamous Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MO22089; 2008-007008-27
Record Dates: First submitted 2009-08-18; First posted 2009-08-19 (Estimated); Results first posted 2016-02-22 (Estimated); Last update posted 2016-02-22 (Estimated); Status verified 2016-01

CONDITIONS: Non-Squamous Non-Small Cell Lung Cancer
MeSH Terms: interventions — Bevacizumab; Cisplatin; Pemetrexed

ARMS (3):
- Part 1 (Experimental)
  Interventions: Drug: bevacizumab [Avastin]; Drug: cisplatin; Drug: pemetrexed
- Part 2A (Experimental)
  Interventions: Drug: bevacizumab [Avastin]
- Part 2B (Active Comparator)
  Interventions: Drug: bevacizumab [Avastin]; Drug: pemetrexed

INTERVENTIONS:
Drug: bevacizumab [Avastin] — 7.5mg/kg iv on day 1 of each 3-week cycle
Drug: cisplatin — 75mg/m2 iv on day 1 of each 3-week cycle
  Arms: Part 1
Drug: pemetrexed — 500mg/m2 iv on day 1 of each 3-week cycle
  Arms: Part 1; Part 2B

SUMMARY:
This open-label study will assess the efficacy and safety of Avastin with or without pemetrexed as maintenance therapy in patients with advanced, metastatic or recurrent non-small cell lung cancer. In Part 1, patients will receive 4 cycles of treatment with Avastin (7.5mg/kg iv) plus cisplatin (75mg/m2 iv) plus pemetrexed (500mg/m2 iv) on day 1 of each 3-week cycle. In Part 2, patients responding to treatment will be randomized to receive further treatment cycles of Avastin (7.5mg/kg iv every 3 weeks) with or without pemetrexed (500mg/m2 iv every 3 weeks). Anticipated time on study treatment is until disease progression. Target sample size is <500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adults >/=18 years of age
* inoperable, locally advanced, metastatic or recurrent non-squamous non-small cell lung cancer (NSCLC)
* at least 1 measurable lesion meeting RECIST criteria
* ECOG performance status 0-2
* adequate hematological, liver and renal function

Exclusion Criteria:

* prior chemotherapy or treatment with another systemic anti-cancer agent
* malignancies other than NSCLC within 5 years prior to randomization, except for adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer, localized prostate cancer or DCIS
* evidence of tumor invading major blood vessels
* current or recent use of aspirin (>325mg/day) or full-dose anticoagulants or thrombolytic agents for therapeutic purposes
* history of haemoptysis >/=grade 2
* clinically significant cardiovascular disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 376 (Actual)
Dates: Start 2009-08; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (82):
- France (24):
  - Béziers
  - Bordeaux
  - Bron
  - Caen
  - Clermont-Ferrand
  - Créteil
  - Gap
  - Gleizé
  - La Source
  - La Tronche
  - Lille
  - Limoges
  - Lyon
  - Marseille
  - Nancy
  - Nîmes
  - Paris
  - Perpignan
  - Pierre-Bénite
  - Reims
  - Saint-Priest-en-Jarez
  - Strasbourg
  - Toulon
  - Tours
- Germany (17):
  - Augsburg
  - Bad Berka
  - Berlin
  - Bonn
  - Ebensfeld
  - Frankfurt
  - Freiburg im Breisgau
  - Gauting
  - Großhansdorf
  - Halle
  - Hamburg
  - Immenhausen
  - Karlsruhe
  - Leipzig
  - Minden
  - München
  - Oldenburg
- Alexandroupoli, Greece
- Italy (8):
  - Lecce, Apulia
  - Napoli, Campania
  - Aviano, Friuli Venezia Giulia
  - Rome, Lazio
  - Novara, Piedmont
  - Sassari, Sardinia
  - Pisa, Tuscany
  - Padua, Veneto
- Netherlands (11):
  - 's-Hertogenbosch
  - Amersfoort
  - Amsterdam
  - Breda
  - Eindhoven
  - Haarlem
  - Nieuwegein
  - Rotterdam
  - Sittard-Geleen
  - The Hague
  - Zaandam
- Russia (5):
  - Balashikha
  - Irkutsk
  - Krasnodar
  - Moscow
  - Saint Petersburg
- South Korea (4):
  - Bundang City
  - Daegu
  - Gyeonggi-do
  - Seoul
- Spain (4):
  - Palma de Mallorca, Balearic Islands
  - Las Palmas de Gran Canaria, Las Palmas
  - Madrid, Madrid
  - San Cristóbal de La Laguna, Tenerife
- Sweden (4):
  - Gävle
  - Linköping
  - Lund
  - Uppsala
- Zurich, Switzerland
- Turkey (Türkiye) (2):
  - Antalya
  - Izmir
- Al Ain City, United Arab Emirates

REFERENCES:
- [Derived] Barlesi F, Scherpereel A, Rittmeyer A, Pazzola A, Ferrer Tur N, Kim JH, Ahn MJ, Aerts JG, Gorbunova V, Vikstrom A, Wong EK, Perez-Moreno P, Mitchell L, Groen HJ. Randomized phase III trial of maintenance bevacizumab with or without pemetrexed after first-line induction with bevacizumab, cisplatin, and pemetrexed in advanced nonsquamous non-small-cell lung cancer: AVAPERL (MO22089). J Clin Oncol. 2013 Aug 20;31(24):3004-11. doi: 10.1200/JCO.2012.42.3749. Epub 2013 Jul 8. PMID 23835708

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 414 participants were screened out of which 38 participants were excluded for not meeting the eligibility criteria, declining to participate, or for other reasons. A total of 376 participants were recruited over an 18-month period across 81 centers in 11 countries from 17 August 2009 to 3 May 2011.
Pre-assignment Details: Of the 376 participants enrolled in this study, 3 participants did not start induction phase treatment.
Groups:
- Induction Treatment Phase: Bevacizumab 7.5 milligram (mg)/ kilogram (kg) + cisplatin 75 mg/m^2 + pemetrexed 500 mg/m^2 was administered intravenously (IV) every 3 weeks. Participants received 4 cycles of induction therapy.
- Bevacizumab Maintenance Treatment (Trt) Arm A: Bevacizumab 7.5 mg/kg was administered IV every 3 weeks until progression of disease, unacceptable toxicity, or withdrawal of consent. The first cycle of maintenance therapy was to be administered a maximum of 4 weeks after the fourth cycle of induction therapy.
- Bevacizumab +Pemetrexed Maintenance Trt Arm B: Bevacizumab 7.5 mg/kg + pemetrexed 500 mg/m^2 was administered IV every 3 weeks until progression of disease, unacceptable toxicity, or withdrawal of consent. Pemetrexed-treated participants received standard supplementation with folic acid orally (350 to 1000 microgram [mcg] daily), vitamin B12 intramuscularly (1000 mcg every 3 cycles), and dexamethasone prophylaxis orally (4 mg twice a day) on Days -1, 1, and 2 of each cycle. The first cycle of maintenance therapy was to be administered a maximum of 4 weeks after the fourth cycle of induction therapy.
Period: Induction Treatment Phase
Arm/Group | Induction Treatment Phase | Bevacizumab Maintenance Treatment (Trt) Arm A | Bevacizumab +Pemetrexed Maintenance Trt Arm B
Started | 376 | 0 | 0
Completed | 253 | 0 | 0
Not Completed | 123 | 0 | 0
Not completed — Withdrawal by Subject | 11 | 0 | 0
Not completed — Death | 77 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Physician Decision | 2 | 0 | 0
Not completed — Didn't meet maintenance phase criteria | 27 | 0 | 0
Not completed — Other Reason | 5 | 0 | 0
Period: Maintenance Treatment Phase
Arm/Group | Induction Treatment Phase | Bevacizumab Maintenance Treatment (Trt) Arm A | Bevacizumab +Pemetrexed Maintenance Trt Arm B
Started | 0 | 125 | 128
Completed | 0 | 77 | 83
Not Completed | 0 | 48 | 45
Not completed — Death | 0 | 42 | 34
Not completed — Investigators decision | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 3 | 8
Not completed — Other reason | 0 | 1 | 3

BASELINE CHARACTERISTICS:
Population: The Intent-to-treat (ITT) population included all the participants that were randomized.
Groups:
- Bevacizumab Maintenance Trt Arm A: Bevacizumab 7.5 mg/kg was administered IV every 3 weeks until progression of disease, unacceptable toxicity, or withdrawal of consent. The first cycle of maintenance therapy had to be administered a maximum of 4 weeks after the fourth cycle of induction therapy.
- Total: Total of all reporting groups
Arm/Group | Bevacizumab Maintenance Trt Arm A | Bevacizumab +Pemetrexed Maintenance Trt Arm B | Total
Number analyzed (Participants) | 125 | 128 | 253
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.5 (8.25) | 59.3 (8.86) | 59.4 (8.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 54 | 109
  Male | 70 | 74 | 144

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival During Maintenance Treatment Phase
Description: Progression free survival (PFS) is defined as the time from randomization to the date of documented disease progression according to Response Evaluation Criteria in Solid Tumors (RECIST v1.1) , or the date of occurrence of a second primary cancer, or date of death from any cause, whichever comes first. Progression is defined using (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, the appearance of new lesions and increase of at least 5 mm in the sum of diameters of target lesions.Tumor assessment was done before Cycle 3, at Cycle 2 of maintenance therapy and every nine weeks thereafter.
Time Frame: Up to 21 months
Population: The ITT population included all the participants that were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Bevacizumab Maintenance Trt Arm A | Bevacizumab +Pemetrexed Maintenance Trt Arm B
Number analyzed (Participants) | 125 | 128
Months | 6.6 [6.0 to 7.8] | 10.2 [9.1 to 11.7]
Statistical Analysis 1: Comparison: Bevacizumab Maintenance Trt Arm A vs Bevacizumab +Pemetrexed Maintenance Trt Arm B; Test type: Superiority or Other; p < 0.001, Log Rank; Hazard Ratio (HR) = 0.50, 95% CI 2-sided [0.37 to 0.69]

2. Secondary Outcome: Overall Survival During Maintenance Treatment Phase
Description: Overall survival (OS) is assessed from the date of first induction treatment until the date of death. Tumor assessment was done before Cycle 3, at Cycle 2 of maintenance therapy and every nine weeks thereafter.
Time Frame: Up to 21 months
Population: The ITT population included all the participants that were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Bevacizumab Maintenance Trt Arm A | Bevacizumab +Pemetrexed Maintenance Trt Arm B
Number analyzed (Participants) | 125 | 128
Months | 15.7 [14.3 to NA] — Data unavailable, as the follow-up time was very short to observe enough survival events. | NA [NA to NA] — Data unavailable, as the follow-up time was very short to observe enough survival events.
Statistical Analysis 1: Comparison: Bevacizumab Maintenance Trt Arm A vs Bevacizumab +Pemetrexed Maintenance Trt Arm B; Test type: Superiority or Other; p = 0.230, Log Rank; Hazard Ratio (HR) = 0.75, 95% CI 2-sided [0.47 to 1.20]

3. Secondary Outcome: Best Overall Response Rate During Maintenance Treatment Phase
Description: The best overall response rate (BORR) is defined as the percentage of participants having achieved confirmed Complete Response (CR) and Partial Response (PR) as the best overall response. CR was defined as complete disappearance of all target lesions and non-target disease. PR was defined as a greater than or equal to (≥) 30% decrease under baseline of the sum of diameters of all target lesions. Stable disease (SD) is defined as steady state of disease with neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD).Tumor assessment was done before Cycle 3, at Cycle 2 of maintenance therapy and every nine weeks thereafter.
Time Frame: Up to 21 months
Population: The ITT population which included all the participants that were randomized.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab Maintenance Trt Arm A | Bevacizumab +Pemetrexed Maintenance Trt Arm B
Number analyzed (Participants) | 125 | 128
percentage of participants
  Partial response (PR) | 50 [40.9 to 59.1] | 55.5 [46.4 to 64.3]
  Stable disease (SD) | 50 [40.9 to 59.1] | 44.5 [35.7 to 53.6]

4. Secondary Outcome: Duration of Response During Maintenance Treatment Phase
Description: Duration of response is defined as the time in months from the initial start of response PR or better to the earlier of documented PD or death due to any cause. Participants who had neither progressed nor died at the date of clinical cutoff, who withdrew from the study, were lost to follow-up, or were without documented disease progression were censored at the date of the last available tumor assessment. The analysis was based on all participants with measurable disease at baseline who achieved response.Tumor assessment was done before Cycle 3, at Cycle 2 of maintenance therapy and every nine weeks thereafter.
Time Frame: Up to 21 months
Population: The ITT population included all the participants that were randomized.Participants available at particular time point for assessment were included in the analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Bevacizumab Maintenance Trt Arm A | Bevacizumab +Pemetrexed Maintenance Trt Arm B
Number analyzed (Participants) | 62 | 71
Months | 5.7 [4.9 to 7.2] | 9.2 [6.8 to 10.4]
Statistical Analysis 1: Comparison: Bevacizumab Maintenance Trt Arm A vs Bevacizumab +Pemetrexed Maintenance Trt Arm B; Test type: Superiority or Other; p = 0.006, Log Rank; Hazard Ratio (HR) = 0.53, 95% CI 2-sided [0.34 to 0.84]

5. Secondary Outcome: Duration of Disease Control During Maintenance Treatment Phase
Description: Duration of disease control is defined as the time in months from randomization to the earlier of documented PD or death due to any cause. Tumor assessment was done before Cycle 3, at Cycle 2 of maintenance therapy and every nine weeks thereafter.
Time Frame: Up to 21 months
Population: The ITT population included all the participants that were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Bevacizumab Maintenance Trt Arm A | Bevacizumab +Pemetrexed Maintenance Trt Arm B
Number analyzed (Participants) | 125 | 128
Months | 4.9 [3.9 to 5.7] | 7.8 [6.8 to 9.7]
Statistical Analysis 1: Comparison: Bevacizumab Maintenance Trt Arm A vs Bevacizumab +Pemetrexed Maintenance Trt Arm B; Test type: Superiority or Other; p < 0.001, Log Rank; Hazard Ratio (HR) = 0.52, 95% CI 2-sided [0.38 to 0.70]

6. Secondary Outcome: Incidence of Adverse Events and Serious Adverse Event
Description: An adverse events (AE) is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not considered related to the medicinal (investigational) product. An serious adverse event (SAE) is any experience that suggests a significant hazard, contraindication, side effect, or precaution.
Time Frame: Up to 21 months
Population: The safety population comprised of all participants who received at least one dose of study medication. Participants who received induction treatment and were not randomised to maintenance treatment are also included in analysis.
Measure: Number; unit: Participants
Groups:
- Bevacizumab Maintenance Trt Arm A: Bevacizumab 7.5 mg/kg was administered IV every 3 weeks until progression of disease, unacceptable toxicity, or withdrawal of consent. Among the 125 participants allocated to Bevacizumab Maintenance Trt Arm A, five participants did not receive treatment so they were excluded from analysis.
- Bevacizumab +Pemetrexed Maintenance Trt Arm B: Bevacizumab 7.5 mg/kg + pemetrexed 500mg/m^2 was administered IV every 3 weeks until progression of disease, unacceptable toxicity, or withdrawal of consent. Among the 128 participants allocated to Bevacizumab +Pemetrexed Maintenance Trt Arm B, three participants did not receive treatment so they were excluded from analysis.
- No Maintenance Trt: A total of 128 participants were not randomized to maintenance therapy because of discontinuations related to an AE, progressive disease, withdrawal of consent, or other reasons. Five participants in Bevacizumab Maintenance Trt Arm A and three in Bevacizumab +Pemetrexed Maintenance Trt Arm B, respectively, did not receive maintenance treatment so they were also included in the not randomized arm.
Arm/Group | Bevacizumab Maintenance Trt Arm A | Bevacizumab +Pemetrexed Maintenance Trt Arm B | No Maintenance Trt
Number analyzed (Participants) | 120 | 125 | 128
Participants
  AE | 116 | 123 | 119
  SAE | 26 | 42 | 70

7. Secondary Outcome: Number of Participants With Marked Laboratory Abnormalities
Description: Marked laboratory abnormalities were defined as those values that were outside the reference range and showed a clinically relevant change from Baseline. The reference range for Platelets was 100-550 (10^9/L), for White blood cells (WBC) was 3.0-18.0 (10^9/L), for Lymphocytes was 0.70-7.60 (10^9/L), and Neutrophil 1.50-9.25 (10^9/L ).
Time Frame: Up to 21 months
Population: as for outcome 6
Measure: Number; unit: Participants
Arm/Group | Bevacizumab Maintenance Trt Arm A | Bevacizumab +Pemetrexed Maintenance Trt Arm B | No Maintenance Trt
Number analyzed (Participants) | 120 | 125 | 128
Participants
  Alanine amino transferase (ALT) | 18 | 26 | 8
  Aspartate amino transferase (AST) | 18 | 26 | 8
  Alkaline phosphatase | 18 | 26 | 8
  Hemoglobin | 28 | 30 | 25
  International normalized ratio (INR) | 1 | 0 | 0
  Lymphocytes | 28 | 30 | 25
  Neutrophils | 28 | 30 | 25
  Platelets | 28 | 30 | 25
  Serum creatinine | 18 | 26 | 8
  WBC | 28 | 30 | 25
  Activated partial thromboplastin time (aPTT) | 1 | 0 | 0

8. Secondary Outcome: Quality of Life
Description: European Organization for Research and Treatment of Cancer Quality-of-Life Questionnaire-Cancer 30 (EORTC QLQ-C30): included functional scales (physical, role, cognitive, emotional, and social), global health status, symptom scales (fatigue, pain, nausea/vomiting) and single items (dyspnoea, appetite loss, insomnia, constipation/diarrhea and financial difficulties). The European Organization for Research and Treatment of Cancer Quality-of-Life Questionnaire-Lung Cancer 13 [EORTC QLQ-LC13]consisted of 1 multi-item scale and 9 single items that assessed the specific symptoms (dyspnea, cough, hemoptysis, and site specific pain), side effects (sore mouth, dysphagia, neuropathy, and alopecia), and pain medication use of lung cancer participants receiving chemotherapy. Scale score range: 0 to 100. Higher symptom score = greater degree of symptom severity. QOL was assessed using Pre-Induction Baseline (Pre-ind BL), Maintenance (MTC), End of study (EOS) cycles.
Time Frame: Up to 21 months
Population: The ITT population included all the participants that were randomized.
Measure: Mean (Standard Deviation); unit: Score on scale
Groups:
- Bevacizumab +Pemetrexed Maintenance Trt Arm B: Bevacizumab 7.5 mg/kg + pemetrexed 500 mg/m^2 was administered IV every 3 weeks until progression of disease, unacceptable toxicity, or withdrawal of consent. Pemetrexed-treated participants received standard supplementation with folic acid orally (350 to 1000 mcg daily), vitamin B12 intramuscularly (1000 mcg every 3 cycles), and dexamethasone prophylaxis orally (4 mg twice a day) on Days -1, 1, and 2 of each cycle. The first cycle of maintenance therapy was to be administered a maximum of 4 weeks after the fourth cycle of induction therapy.
Arm/Group | Bevacizumab Maintenance Trt Arm A | Bevacizumab +Pemetrexed Maintenance Trt Arm B
Number analyzed (Participants) | 125 | 128
Score on scale
  [Pre-ind BL] Global Health Status Scale n=116,121 | 57.9 (23.90) | 59.7 (21.74)
  [Pre-ind BL] Physical Functional Scale (n=118,121) | 74.8 (23.69) | 79.4 (18.09)
  [Pre-ind BL] Role Functional Scale (n=118,121) | 68.4 (32.50) | 71.1 (28.28)
  [Pre-ind BL] Emotional Functional Scale n=117,121 | 71.7 (21.93) | 69.8 (21.97)
  [Pre-ind BL] Cognitive Functional Scale n=117,121 | 86.0 (21.55) | 88.0 (16.70)
  [Pre-ind BL]] Social Functional Scale (n=116,120) | 79.3 (25.60) | 78.7 (26.10)
  [Pre-ind BL] Fatigue Symptom Scale (n=118,121) | 33.3 (27.18) | 31.5 (21.73)
  [Pre-ind BL] Nausea & Vomiting Scale n=118,121 | 7.2 (17.50) | 4.3 (12.46)
  [Pre-ind BL] Pain Symptom Scale (n=118,121) | 36.7 (31.92) | 24.7 (26.88)
  [Pre-ind BL] Dyspnea Symptom Scale (n=118,121) | 29.7 (30.75) | 30.6 (29.69)
  [Pre-ind BL] Insomnia Symptom Scale n=118,121 | 33.3 (34.59) | 33.9 (30.42)
  [Pre-ind BL] Appetite Loss Symptom Scale n=118,121 | 19.2 (30.01) | 18.7 (29.15)
  [Pre-ind BL]] Constipation Symptom Scale n=118,121 | 18.6 (30.68) | 9.1 (20.18)
  [Pre-ind BL] Diarrhea Symptom Scale (n=117,121) | 7.1 (17.96) | 5.2 (14.91)
  [Pre-ind BL]Financial Difficulties Scale n=114,120 | 17.3 (30.48) | 17.2 (29.62)
  [MTC Cycle 3]Global Health Status (n=69,87) | 63.3 (20.02) | 58.6 (19.71)
  [MTC Cycle 3]Physical Functional Scale (n=69,87) | 77.1 (20.72) | 76.0 (20.37)
  [MTC Cycle 3]Role Functional Scale (n=69,87) | 74.2 (27.79) | 69.9 (28.51)
  [MTC Cycle 3]Emotional Functional Scale (n=69,87) | 82.5 (19.86) | 78.4 (18.48)
  [MTC Cycle 3]Cognitive Functional Scale (n=69,87) | 84.3 (23.20) | 82.6 (19.17)
  [MTC Cycle 3]Social Functional Scale (n=69,87) | 82.1 (25.62) | 73.0 (24.28)
  [MTC Cycle 3]Fatigue Symptom Scale (n=69,87) | 32.1 (22.88) | 34.5 (21.50)
  [MTC Cycle 3]Nausea and Vomiting Scale (n=69,87) | 7.2 (16.78) | 8.8 (12.92)
  [MTC Cycle 3]Pain Symptom Scale (n=69,87) | 23.9 (27.64) | 17.4 (21.85)
  [MTC Cycle 3]Dyspnea Symptom Scale (n=69,87) | 26.1 (27.93) | 29.9 (26.91)
  MTC Cycle 3]Appetite Loss Symptom Scale (n=69,87) | 13.5 (22.37) | 18.4 (25.80)
  [MTC Cycle 3]Insomnia Symptom Scale (n=69,87) | 19.3 (24.53) | 19.5 (25.19)
  [MTC Cycle 3]Constipation Symptom Scale (n=69,87) | 10.1 (19.22) | 11.1 (20.12)
  [MTC Cycle 3]Diarrhea Symptom Scale (n=69,87) | 3.4 (12.97) | 5.7 (14.56)
  [MTC Cycle 3]Financial Difficulties Scale (n=68,86 | 18.1 (27.88) | 19.4 (26.30)
  [MTC Cycle 5] Global Health Status (n=51,77) | 63.2 (20.36) | 62.9 (18.81)
  [MTC Cycle 5] Physical Functional Scale (n=51,77) | 78.7 (21.29) | 78.4 (15.45)
  [MTC Cycle 5] Role Functional Scale (n=51,77) | 74.5 (31.15) | 68.8 (27.08)
  [MTC Cycle 5] Emotional Functional Scale (n=51,77) | 78.8 (23.76) | 78.7 (20.96)
  [MTC Cycle 5] Cognitive Functional Scale (n=51,77) | 81.0 (26.04) | 84.6 (18.09)
  [MTC Cycle 5] Social Functional Scale (n=51,77) | 85.3 (22.52) | 77.9 (22.85)
  [MTC Cycle 5] Fatigue Symptom Scale (n=51,77) | 32.2 (23.01) | 34.5 (22.12)
  [MTC Cycle 5] Nausea and Vomiting Scale (n=51,77) | 9.2 (18.05) | 10.0 (20.10)
  [MTC Cycle 5] Pain Symptom Scale (n=51,77) | 23.5 (26.28) | 20.1 (25.27)
  [MTC Cycle 5] Dyspnea Symptom Scale (n=51,77) | 25.5 (27.96) | 35.9 (30.95)
  [MTC Cycle 5] Insomnia Symptom Scale( n=51,77) | 21.6 (28.92) | 22.1 (27.36)
  MTC Cycle 5] Appetite Loss Symptom Scale (n=51,77) | 10.5 (19.43) | 19.9 (26.63)
  [MTC Cycle 5] Constipation Symptom Scale (n=51,77) | 9.2 (20.09) | 17.3 (29.42)
  [MTC Cycle 5] Diarrhea Symptom Scale (n=51,77) | 10.5 (20.54) | 2.6 (8.99)
  [MTC Cycle 5] Financial Difficulties Scale n=50,77 | 16.0 (28.76) | 17.7 (23.31)
  [MTC Cycle 7] Global Health Status Scale (n=38,64) | 61.2 (21.69) | 61.3 (19.55)
  [MTC Cycle 7] Physical Functional Scale (n=38,64) | 75.6 (21.49) | 74.7 (19.38)
  [MTC Cycle 7]Role Functional Scale (n=38,64) | 76.8 (24.97) | 70.8 (28.79)
  [MTC Cycle 7]Emotional Functional Scale (n=38,64) | 81.6 (22.27) | 77.5 (18.64)
  [MTC Cycle 7]Cognitive Functional Scale (n=38,64) | 77.2 (27.51) | 81.0 (18.98)
  [MTC Cycle 7]Social Functional Scale (n=38,64) | 82.9 (24.35) | 72.1 (28.65)
  [MTC Cycle 7]Fatigue Symptom Scale (n=38,64) | 32.3 (22.07) | 33.7 (24.72)
  [MTC Cycle 7]Nausea & Vomiting Scale (n=38,64) | 8.3 (18.88) | 9.6 (16.48)
  [MTC Cycle 7]Pain Symptom Scale (n=38,64) | 21.5 (23.86) | 19.8 (23.55)
  [MTC Cycle 7]Dyspnea Symptom Scale (n=38,64) | 28.1 (26.31) | 37 (32.59)
  [MTC Cycle 7]Insomnia Symptom Scale (n=38,64) | 16.7 (26.57) | 28.6 (30.21)
  [MTC Cycle 7]Appetite Loss Scale (n=38,64) | 12.3 (21.11) | 21.4 (29.32)
  [MTC Cycle 7]Constipation Symptom Scale (n=38,64) | 14 (28.61) | 17.2 (24.48)
  [MTC Cycle 7]Diarrhea Symptom Scale (n=38,64) | 8.8 (20.04) | 8.9 (21.61)
  [MTC Cycle 7]Financial Difficulties Scale n=38,64 | 14.0 (24.05) | 20.3 (27.61)
  [MTC Cycle 9 ]Global Health Status Scale (n=33,50) | 60.6 (18.67) | 61.2 (17.71)
  [MTC Cycle 9 ]Physical Functional Scale (n=33,50) | 80.8 (20.53) | 74.9 (19.54)
  [MTC Cycle 9 ]Role Functional Scale (n=33,50) | 75.8 (24.33) | 69.7 (28.51)
  [MTC Cycle 9 ]Emotional Functional Scale (n=33,50) | 82.3 (18.61) | 75 (22.46)
  [MTC Cycle 9 ]Cognitive Functional Scale (n=33,50) | 83.3 (20.41) | 81.7 (19.99)
  [MTC Cycle 9 ]Social Functional Scale (n=33,50) | 83.8 (24.47) | 71.7 (26.78)
  [MTC Cycle 9 ]Fatigue Symptom Scale (n=33,50) | 28.3 (24.07) | 35.1 (25.03)
  [MTC Cycle 9 ]Nausea & Vomiting Symptom (n=33,50) | 5.1 (12.14) | 12.0 (20.77)
  [MTC Cycle 9 ]Pain Symptom Scale (n=33,50) | 25.8 (30.93) | 18.7 (21.47)
  [MTC Cycle 9 ]Dyspnea Symptom Scale (n=32,50) | 25.0 (25.40) | 35.3 (27.28)
  [MTC Cycle 9 ]Insomnia Symptom Scale (n=33,49) | 23.2 (26.98) | 30.6 (33.91)
  [MTC Cycle 9 ]Appetite Loss Scale (n=33,50) | 10.1 (19.52) | 23.3 (29.55)
  [MTC Cycle 9 ]Constipation Symptom Scale (n=33,50) | 13.1 (24.92) | 16.0 (25.41)
  [MTC Cycle 9 ]Diarrhea Symptom Scale (n=33,50) | 7.1 (20) | 7.3 (18.18)
  [MTC Cycle 9]Financial Difficulties Scale n=33,50 | 15.2 (23.70) | 22.0 (27.45)
  [MTC Cycle 11 ] Global Health Status Scale n=25,37 | 57.7 (18.93) | 59.9 (21.41)
  [MTC Cycle 11 ]Physical Functional Scale (n=25,37) | 79.2 (16.48) | 81.1 (17.81)
  [MTC Cycle 11 ]Role Functional Scale (n=25,37) | 77.3 (18.56) | 73.9 (27.37)
  [MTC Cycle 11 ]Emotional Functional Scale n=25,37 | 78.3 (19.09) | 80.0 (19.88)
  [MTC Cycle 11 ]Cognitive Functional Scale n=25,37 | 81.3 (26.49) | 84.2 (17.10)
  [MTC Cycle 11 ]Social Functional Scale (n=25,37) | 84.7 (19.20) | 77.9 (27.51)
  [MTC Cycle 11 ]Fatigue Symptom Scale (n=25,37) | 32.4 (22.20) | 31.2 (20.92)
  [MTC Cycle 11 ]Nausea & Vomiting Scale (n=25,37) | 6.7 (15.96) | 9.5 (18.23)
  [MTC Cycle 11 ]Pain Symptom Scale (n=25,37) | 29.3 (28.98) | 19.8 (27.45)
  [MTC Cycle 11 ]Dyspnea Symptom Scale (n=25,37) | 30.7 (16.44) | 28.8 (27.40)
  [MTC Cycle 11 ]Insomnia Symptom Scale (n=25,37) | 20.0 (23.57) | 18.9 (26.69)
  [MTC Cycle 11 ]Appetite Loss Scale (n=25,37) | 9.3 (20.46) | 18 (26.75)
  MTC Cycle 11 ]Constipation Symptom Scale( n=25,37) | 6.7 (13.61) | 17.1 (24.37)
  [MTC Cycle 11 ]Diarrhea Symptom Scale ( n=25,37) | 1.3 (6.67) | 7.2 (15.98)
  [MTC Cycle 11]Financial Difficulties Scale n=24,37 | 15.3 (25.97) | 18.0 (26.75)
  [EOS]Global Health Status Scale (n=123,127) | 55.1 (20.62) | 57.2 (20.01)
  [EOS]Physical Functional Scale (n=125,127) | 70.2 (23.49) | 72.5 (22.06)
  [EOS]Role Functional Scale (n=125,127) | 63.5 (32.43) | 64.3 (29.68)
  [EOS]Emotional Functional Scale (n=124,127) | 74.4 (21.36) | 77.3 (20.20)
  [EOS]Cognitive Functional Scale ( n=124,127) | 79.3 (24.91) | 83.5 (19.30)
  [EOS]Social Functional Scale (n=124,127) | 73.3 (29.28) | 72.6 (27.90)
  [EOS]Fatigue Symptom Scale (n=125,127) | 41.0 (26.42) | 37.6 (23.80)
  [EOS]Nausea & Vomiting Scale (n=125,127) | 14.4 (23.70) | 12.3 (20.70)
  [EOS]Pain Symptom Scale (n=125,127) | 30.4 (30.31) | 21.1 (25.58)
  [EOS]Dyspnea Symptom Scale (n=124,127) | 31.5 (29.85) | 34.1 (29.83)
  [EOS]Insomnia Symptom Scale( n=125,127) | 27.2 (26.57) | 22.6 (28.45)
  [EOS]Appetite Loss Symptom Scale (n=125,127) | 26.9 (31.31) | 26.0 (30.26)
  [EOS]Constipation Symptom Scale (n=125,127) | 17.6 (25.60) | 12.1 (21.28)
  [EOS]Diarrhea Symptom Scale(n=124,127) | 9.7 (20.72) | 6.8 (15.34)
  [EOS]Financial Difficulties Scale (n=123,126) | 16.8 (27.45) | 16.9 (27.24)

ADVERSE EVENTS:
Time Frame: Up to 21 months (throughout the study)
Description: Serious adverse events and non-serious adverse events are reported in Safety Analysis Set, which consists of all participants who received at least one dose of study medication and had a safety assessment performed post baseline.
Groups:
- No Maintenance Treatment: A total of 128 participants were not randomized to maintenance therapy because of discontinuations related to an AE, progressive disease, withdrawal of consent, or other reasons. Five participants in Bevacizumab Maintenance Trt Arm A and three in Bevacizumab +Pemetrexed Maintenance Trt Arm B, respectively, did not receive maintenance treatment so they were also included in the not randomized arm..
- Maintenance Treatment Arm A: Bevacizumab 7.5 mg/kg was administered IV every 3 weeks until progression of disease, unacceptable toxicity, or withdrawal of consent. Among the 125 participants allocated to Bevacizumab Maintenance Trt Arm A, five participants did not receive treatment so they were excluded from analysis
- Maintenance Treatment Arm B: Bevacizumab 7.5 mg/kg + pemetrexed 500mg/m^2 was administered IV every 3 weeks until progression of disease, unacceptable toxicity, or withdrawal of consent. Among the 128 participants allocated to Bevacizumab +Pemetrexed Maintenance Trt Arm B, three participants did not receive treatment so they were excluded from analysis..
Arm/Group | No Maintenance Treatment | Maintenance Treatment Arm A | Maintenance Treatment Arm B
Serious Adverse Events (participants affected / at risk) | 70/128 | 26/120 | 42/125
Other Adverse Events (participants affected / at risk) | 105/128 | 115/120 | 120/125
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | No Maintenance Treatment (N=128) | Maintenance Treatment Arm A (N=120) | Maintenance Treatment Arm B (N=125)
Pneumonia (Infections and infestations) | 3 | 1 | 7
Anal abscess (Infections and infestations) | 1 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 1
Device related infection (Infections and infestations) | 0 | 1 | 1
Sepsis (Infections and infestations) | 2 | 0 | 0
Abscess limb (Infections and infestations) | 1 | 0 | 0
Clostridial infection (Infections and infestations) | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 1
Gastroenteritis norovirus (Infections and infestations) | 0 | 0 | 1
Intervertebral discitis (Infections and infestations) | 0 | 1 | 0
Lung infection (Infections and infestations) | 0 | 0 | 1
Oesophageal candidiasis (Infections and infestations) | 1 | 0 | 0
Post procedural infection (Infections and infestations) | 1 | 0 | 0
Pulmonary sepsis (Infections and infestations) | 0 | 0 | 1
Scrub typhus (Infections and infestations) | 0 | 0 | 1
Septic shock (Infections and infestations) | 1 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 9 | 3 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Bronchopleural fistula (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 2 | 2
Nausea (Gastrointestinal disorders) | 0 | 2 | 3
Vomiting (Gastrointestinal disorders) | 1 | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 1 | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal toxicity (Gastrointestinal disorders) | 1 | 0 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 1 | 0 | 0
Oesophageal perforation (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Tongue oedema (Gastrointestinal disorders) | 0 | 0 | 1
General physical health deterioration (General disorders) | 3 | 1 | 0
Asthenia (General disorders) | 1 | 1 | 1
Death (General disorders) | 2 | 0 | 1
Malaise (General disorders) | 2 | 0 | 1
Pain (General disorders) | 1 | 0 | 1
Pyrexia (General disorders) | 1 | 0 | 1
Sudden death (General disorders) | 2 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0
Haemorrhagic cyst (General disorders) | 0 | 1 | 0
Hyperthermia (General disorders) | 0 | 1 | 0
Impaired healing (General disorders) | 0 | 0 | 1
Mucosal inflammation (General disorders) | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 4 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 7 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 1
Pancytopenia (Blood and lymphatic system disorders) | 1 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0 | 0
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 3 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 3 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypercreatininaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 2 | 0
Thrombophlebitis (Vascular disorders) | 1 | 0 | 1
Embolism arterial (Vascular disorders) | 1 | 0 | 0
Embolism venous (Vascular disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 1 | 0
Iliac artery embolism (Vascular disorders) | 1 | 0 | 0
Ischaemia (Vascular disorders) | 1 | 0 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0 | 0
Peripheral ischaemia (Vascular disorders) | 0 | 0 | 1
Thrombophlebitis superficial (Vascular disorders) | 0 | 0 | 1
Vasculitis necrotising (Vascular disorders) | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 2
Cerebral haemorrhage (Nervous system disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 1
Nervous system disorder (Nervous system disorders) | 0 | 0 | 1
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 1 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0
Viith nerve paralysis (Nervous system disorders) | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 4 | 0 | 2
Renal failure acute (Renal and urinary disorders) | 2 | 0 | 0
Renal impairment (Renal and urinary disorders) | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 1
Cardiac asthma (Cardiac disorders) | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 1 | 0 | 0
Cardiogenic shock (Cardiac disorders) | 1 | 0 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0 | 0
General physical condition abnormal (Investigations) | 2 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 0
White blood cell count decreased (Investigations) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0
Hepatic vein thrombosis (Hepatobiliary disorders) | 1 | 0 | 0
Hepatotoxicity (Hepatobiliary disorders) | 1 | 0 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Respiratory fume inhalation disorder (Injury, poisoning and procedural complications) | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 0 | 1
Vitreous detachment (Eye disorders) | 0 | 0 | 1
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | No Maintenance Treatment (N=128) | Maintenance Treatment Arm A (N=120) | Maintenance Treatment Arm B (N=125)
Nausea (Gastrointestinal disorders) | 47 | 73 | 77
Vomiting (Gastrointestinal disorders) | 21 | 28 | 33
Constipation (Gastrointestinal disorders) | 21 | 33 | 32
Diarrhoea (Gastrointestinal disorders) | 22 | 16 | 35
Abdominal pain upper (Gastrointestinal disorders) | 8 | 8 | 11
Abdominal pain (Gastrointestinal disorders) | 4 | 5 | 8
Stomatitis (Gastrointestinal disorders) | 3 | 6 | 8
Dry mouth (Gastrointestinal disorders) | 2 | 1 | 7
Asthenia (General disorders) | 25 | 42 | 31
Fatigue (General disorders) | 22 | 22 | 40
Chest pain (General disorders) | 11 | 15 | 15
Mucosal inflammation (General disorders) | 12 | 7 | 15
Oedema peripheral (General disorders) | 7 | 4 | 19
Pyrexia (General disorders) | 8 | 6 | 16
Cough (Respiratory, thoracic and mediastinal disorders) | 19 | 27 | 27
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 17 | 26 | 24
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12 | 21 | 26
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 5 | 7 | 8
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 6 | 4
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 9
Neutropenia (Blood and lymphatic system disorders) | 5 | 26 | 26
Anaemia (Blood and lymphatic system disorders) | 17 | 20 | 21
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 8 | 3
Leukopenia (Blood and lymphatic system disorders) | 2 | 6 | 8
Hypertension (Vascular disorders) | 23 | 43 | 55
Headache (Nervous system disorders) | 10 | 19 | 26
Dizziness (Nervous system disorders) | 9 | 7 | 11
Paraesthesia (Nervous system disorders) | 3 | 4 | 11
Dysgeusia (Nervous system disorders) | 7 | 6 | 7
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 3 | 9
Back pain (Musculoskeletal and connective tissue disorders) | 12 | 11 | 13
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 14 | 11
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 11 | 11
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 5 | 11
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 11 | 2
Decreased appetite (Metabolism and nutrition disorders) | 24 | 23 | 32
Hyperglycaemia (Metabolism and nutrition disorders) | 7 | 2 | 8
Weight decreased (Investigations) | 16 | 7 | 8
Blood creatinine increased (Investigations) | 1 | 6 | 11
Haemoglobin decreased (Investigations) | 7 | 0 | 7
Alanine aminotransferase increased (Investigations) | 0 | 3 | 7
Nasopharyngitis (Infections and infestations) | 1 | 8 | 19
Bronchitis (Infections and infestations) | 1 | 8 | 7
Urinary tract infection (Infections and infestations) | 5 | 3 | 7
Alopecia (Skin and subcutaneous tissue disorders) | 8 | 11 | 20
Rash (Skin and subcutaneous tissue disorders) | 0 | 6 | 7
Proteinuria (Renal and urinary disorders) | 4 | 8 | 10
Renal impairment (Renal and urinary disorders) | 3 | 6 | 7
Lacrimation increased (Eye disorders) | 4 | 3 | 16
Conjunctivitis (Eye disorders) | 0 | 6 | 5
Insomnia (Psychiatric disorders) | 4 | 9 | 9
Tachycardia (Cardiac disorders) | 4 | 6 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.